CLINICAL TRIAL: NCT06477159
Title: Pancreatic Enzyme Replacement Therapy for Acute Pancreatitis-Associated Exocrine Pancreatic Insufficiency: the PERT-AP Trial
Brief Title: Pancreatic Enzyme Replacement Therapy for Acute Pancreatitis-Associated Exocrine Pancreatic Insufficiency
Acronym: PERT-AP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Pittsburgh (Other); University of Illinois Chicago (Unknown); University of Southern California (Other); New York University (Other); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0394
Record Dates: First submitted 2024-05-13; First posted 2024-06-27 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pancrelipase (Experimental): Pancrelipase (CREON) capsules taken orally with food, at a dose 36,000 units with snacks and 72,000 units with meals, for a total of 6 months (180 days)
  Interventions: Drug: Pancrelipase Capsules

INTERVENTIONS:
Drug: Pancrelipase Capsules — Treatment with Pancreatic Enzyme Replacement Therapy
  Other Names: CREON

SUMMARY:
This study aims to evaluate if a 6-month course of pancrelipase (CREON) treatment improves symptoms of exocrine pancreatic insufficiency (EPI) after an attack of acute pancreatitis. Diagnosis of EPI is measured by a fecal elastase value of <200, and patients must have a qualifying symptom burden based on the EPI symptom tracker survey. Blood and stool will be analyzed as part of this study, and other surveys of health status will be used to track improvement of symptoms.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, single-arm study of pancrelipase (CREON) in eligible outpatient adults following an episode of acute pancreatitis. Following study eligibility evaluation and informed consent, patients will complete a 7-day run-in period without any pancreatic enzyme replacement therapy and complete baseline questionnaires and assessments, followed by a 180-day treatment period with pancrelipase. The study will end after a final 30 day-post pancrelipase treatment observation period during which safety events will be collected, and EPI symptom burden as well as stool frequency and consistency will be assessed as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of age 18 or older, able to provide informed consent and follow all study procedures.
2. Stable outpatient up to 12 months following an acute pancreatitis episode and has EPI based on an FE-1 < 200 µg/g stool obtained within 3 months prior to baseline assessment (Visit 2).
3. Score of equal or greater 0.6 on the EPI symptom tracker at baseline Visit 2.
4. Must be off PERT (including prescription and non-prescription enzymes) for 7 days prior to baseline Visit 2.
5. Must have fully completed the terminal intervention for necrotizing pancreatitis (surgical or endoscopic necrosectomy or percutaneous drainage).
6. Have a Body Weight between 40 and 120 kg (amounts to 600-1800 LU/meal pancrelipase starting dose of pancrelipase).
7. Women of childbearing potential must have a negative urine pregnancy test at Study Day 1 and practicing at least one protocol specified method of birth control (Section 5.2.4), starting at Study Day 1 through 30 days after last dose of pancrelipase.
8. Females of non-childbearing potential (either postmenopausal or permanently surgically sterile as defined:

   * Age > 55 years with no menses for 12 or more months without an alternative medical cause.
   * Age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 IU/L.

OR

* Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

do not require pregnancy testing.

Exclusion Criteria:

1. Acute pancreatitis episode due to a pancreatic cystic neoplasm, trauma, or surgery. Post-ERCP acute pancreatitis patients can be enrolled.
2. History of definite chronic pancreatitis defined by APA Chronic Pancreatitis Guideline.1
3. Pancreas malignancy or other active malignancies requiring systemic treatment; treated basal cell carcinoma, and treated in-situ cervical cancer can be included.
4. Enteropathies, and gastroenteritis that may affect FE-1 levels, e.g., Inflammatory bowel disease, Celiac Disease, viral-, bacterial-, fungal-, or parasitic gastroenteritis.
5. Gastroparesis.
6. Confirmed or suspected cystic tumor associated with main pancreatic duct dilation or believed to be the cause of AP (in the site-PI's judgment).
7. Prior pancreatic surgery or GI tract surgery affecting the upper GI tract including but not limited to gastric bypass surgery, total pancreatectomy.
8. Pregnancy or breast feeding.
9. Patients with life expectancy of less than 6 months due to advanced chronic conditions, such as congestive heart failure or chronic obstructive pulmonary disease, or other conditions which preclude study participation by judgement of the investigator.
10. Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported EPI Symptoms - Short Term | 30 days
  Determine the patient-reported change in total Exocrine Pancreatic Insufficiency (EPI) symptom score as measured by the EPI Symptom Tracker from baseline to 30 days of pancrelipase treatment; scored from 0 - 3, 0 being no symptoms and 3 being worst possible symptoms.

SECONDARY OUTCOMES:
Patient-Reported EPI Symptoms - LongTerm | 180 days
  Determine the patient-reported change in total Exocrine Pancreatic Insufficiency (EPI)symptom score as measured by the EPI Symptom Tracker from baseline to the end of pancrelipase treatment (180 days); scored from 0 - 3, 0 being no symptoms and 3 being worst possible symptoms.
Change in Stool Frequency | 180 days
  Record changes in stool frequency from baseline to 30 days and from baseline to the end of pancrelipase treatment (180 days)
Change in Stool Consistency | 180 days
  Record change in stool consistency from baseline to 30 days and from baseline to the end of pancrelipase treatment
Change in Depression Score | 180 days
  Change in depression score assessed by the Patient Health Questionnaire (PHQ-9) from baseline to 30 days and from baseline to end of pancrelipase treatment; scores range from 0 - 27, with a higher score meaning worse depression symptoms
Change in SF-12 Health Score | 180 days
  Change in self-assessment of health status as assessed by the 12-Item Short Form Survey (SF-12) from baseline to 30 days and from baseline to end of pancrelipase treatment (180 days); form is not numerically scored
Change in Global Health Score | 180 days
  Change in Global Health score assessed by the Global Health (PROMIS) Questionnaire. Each question is scored 1 - 5, with high values indicating better health status in the first part of the form, and high values indicating poor health status in the latter part of the form; also included is a 0-10 average pain scale.
Medication Adherence | 180 days
  Medication adherence assessed by pill count and the Morisky Medication Adherence Scale (MMAS-8) from baseline to 30 days of pancrelipase treatment and from 30 days to end of pancrelipase treatment (180 days); A score below 6 indicates low adherence, and a score of 8 high adherence. Scale ranges from 0 - 8.
Change in Nutrition Biomarkers - Vitamin D | 180 days
  Change in serum nutrition biomarker Vitamin D (ng/mL)
Change in Nutrition Biomarkers - Retinol Binding Protein | 180 days
  Change in serum nutrition biomarker Retinol Binding Protein (mg/dL)
Change in Nutrition Biomarkers - Pre-albumin | 180 days
  Change in serum nutrition biomarker Pre-albumin (mg/dL)
Change in Nutrition Biomarkers - Albumin | 180 days
  Change in serum nutrition biomarker Albumin (g/dL)

OTHER OUTCOMES:
Frequency, Type, and Severity of Adverse Events | 210 days
  Evaluate the frequency, severity, and causality of adverse events (AEs), treatment emergent AEs (TEAEs), and serious AEs (SAEs); Descriptive assessment of safety and tolerability using FAS set with AEs collected from time of consent to 30 days after end of pancrelipase treatment
Patient-Reported EPI Symptoms - Post-Treatment | 210 days
  Change in total Exocrine Pancreatic Insufficiency (EPI) symptom score as measured by the EPI Symptom Tracker from end of pancrelipase treatment to end of 30-day follow-up period; scored from 0 - 3, 0 being no symptoms and 3 being worst possible symptoms.
Change in Stool Frequency | 210 days
  Change in stool frequency from end of pancrelipase treatment to end of 30-day follow-up period
Change in Stool Consistency | 210 days
  Change in stool consistency from end of pancrelipase treatment to end of 30-day follow-up period

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Southern California, Los Angeles, California
  - University of Illinois Chicago, Chicago, Illinois
  - New York University Langone Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided